CLINICAL TRIAL: NCT04590040
Title: Randomized Non-inferiority Trial of Nano-hydroxyapatite-Containing Toothpastes for Relief of Dentin Hypersensitivity
Brief Title: Trial of Nano-hydroxyapatite-Containing Toothpastes for Relief of Dentin Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Sangi Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Bennett Amaechi, Professor and Director of Cariology, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC20190535H
Record Dates: First submitted 2020-10-03; First posted 2020-10-19 (Actual); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Toothpaste 1 (Active Comparator): Toothpaste 3 containing 5% potassium nitrate (KNO3) will be used by subjects to brush their teeth twice daily for 3 minutes in the morning and before bed each night using a 1 inch strip of toothpaste on a soft-bristled toothbrush.
  Interventions: Device: 5% KNO3 toothpaste
- Toothpaste 2 (Active Comparator): Toothpaste 2 containing 15% nano-HAP will be used by subjects to brush their teeth twice daily for 3 minutes in the morning and before bed each night using a 1 inch strip of toothpaste on a soft-bristled toothbrush.
  Interventions: Device: 15% nano-HAP toothpaste
- Toothpaste 3 (Placebo Comparator): Toothpaste 1 containing 0% nano-hydroxyapatite (HAP) will be used by subjects to brush their teeth twice daily for 3 minutes in the morning and before bed each night using a 1 inch strip of toothpaste on a soft-bristled toothbrush.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — 0% nano-HAP toothpaste
  Other Names: Placebo toothpaste
  Arms: Toothpaste 3
Device: 15% nano-HAP toothpaste — Toothpaste with identical base formulation as the placebo containing 15% nano-HAP
  Other Names: 15 % nano-Hydroxyapatite toothpaste
  Arms: Toothpaste 2
Device: 5% KNO3 toothpaste — Toothpaste with identical base formulation as the placebo containing 5% KNO3
  Other Names: 5% Potassium Nitrate Toothpaste
  Arms: Toothpaste 1

SUMMARY:
Subjects will be enrolled into 3 balanced groups each using a different strength toothpaste. Dental hypersensitivity (DHS) will be assessed at study start, midway and study end.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, placebo-and positive-controlled, stratified parallel group clinical trial. The three groups will be randomly assigned to use one of three test toothpastes having an identical base formulation but containing respectively either 0% nano-hydroxyapatite (HAP) (placebo), 15% nano-HAP or 5% KNO3 (positive control). All dental examinations for data collection will be conducted by the same Clinical Examiner.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the age of 20 and 80 years, of any socio-economic status
* Diagnosed as having DHS, i.e. having at least one sensitive tooth with demonstrated cervical erosion/abrasion or gingival recession
* Showing a sensitivity response to both tactile and cold air stimulus delivered by a Yeaple probe and a one-second blast of cold air respectively
* Patients must be reliable, cooperative and of adequate intelligence to read and understand the rating scales and other study instructions
* Patients must be able to read, comprehend, and sign the informed consent form
* The teeth and sites to be tested should be on the buccal/labial surfaces of incisors, canines, premolars or molars where the affected sites are accessible
* Teeth selected for testing should have a plaque index of ≤ 2

Exclusion Criteria:

* The sensitive tooth is associated with concomitant oral pain due to any other condition such as soft-tissue lesions, tooth-ache ascribable to dental caries, tooth fracture, or cracked tooth syndrome, or pain due to other surgical procedures or injuries.
* The sensitive tooth is associated with a periodontal abscess as diagnosed from an X-ray or clinical examination of the tooth
* The sensitive tooth is associated with mobility >1
* The sensitive tooth is associated with gum pain from gingivitis, occlusal trauma, thermal or chemical burns
* Patients having pain from periodontal-related causes but not DHS
* Previous professional desensitizing treatment
* Patients using medication which could interfere with the perception of pain
* Medical histories marked by chronic use of anti-inflammatory agents, daily analgesics, anticonvulsants, antihistamines, antidepressants, sedatives and/or other psychotropic drugs
* Pregnancy or breastfeeding
* Allergies and idiosyncratic responses to toothpaste ingredients
* Eating disorders or conditions associated with vomiting
* Systemic conditions that are etiologic or predisposing to DHS
* Excessive dietary or environmental exposure to acids
* The sensitive tooth was restored in the preceding three months
* The sensitive tooth is an abutment tooth for fixed or removable prostheses
* The sensitive tooth has extensive restoration or restorations extending into the test area
* Patients below 20 years or above 80 years of age
* Smokers

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bennett T Amaechi, BDS, MS, PhD, Principal Investigator — University of Texas Health at San Antonio
Locations (1):
- School of Dentistry, University of Texas Health Science Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared as de-identified data as summary results reported in ClinicalTrials.gov and in journal publication.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available at study completion

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were consented and enrolled, then for one month there was a washout period. Baseline characteristic measurements were taken prior to washout for both Cold Air Sensitivity and Tactile Stimulus.
Groups:
- Toothpaste 1: Toothpaste 1 containing 0% nano-hydroxyapatite (HAP) will be used by subjects to brush their teeth twice daily for 3 minutes in the morning and before bed each night using a 1 inch strip of toothpaste on a soft-bristled toothbrush.
  Placebo: 0% nano-HAP toothpaste
- Toothpaste 3: Toothpaste 3 containing 5% potassium nitrate (KNO3) will be used by subjects to brush their teeth twice daily for 3 minutes in the morning and before bed each night using a 1 inch strip of toothpaste on a soft-bristled toothbrush.
  5% KNO3 toothpaste: Toothpaste with identical base formulation as the placebo containing 5% KNO3
Period: Washout Period
Arm/Group | Toothpaste 1 | Toothpaste 2 | Toothpaste 3
Started | 64 | 64 | 64
Completed | 64 | 64 | 64
Not Completed | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Toothpaste 1 | Toothpaste 2 | Toothpaste 3
Started | 64 | 64 | 64
Completed | 62 | 59 | 62
Not Completed | 2 | 5 | 2
Not completed — Lost to Follow-up | 2 | 5 | 0
Not completed — Physician Decision | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Toothpaste 1 | Toothpaste 2 | Toothpaste 3 | Total
Number analyzed (Participants) | 62 | 59 | 62 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (16) | 47 (16) | 50 (14) | 48 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 43 | 43 | 130
  Male | 18 | 16 | 19 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 15 | 4 | 12 | 31
  Black (not Hispanic) | 3 | 2 | 1 | 6
  Hispanic | 30 | 28 | 26 | 84
  White (not Hispanic) | 14 | 25 | 23 | 62
Region of Enrollment [Number; unit: participants]
  United States | 62 | 59 | 62 | 183
Cold Air Sensitivity (VAS) [Mean (Standard Deviation); unit: units on a scale] — Tooth sensitivity was measured using a Cold Air Stimulus. When being assessed, participants rated their perception of the pain/discomfort experienced when cold air was directed at the exposed root of each tooth by marking a single vertical line on a Visual Analogue Scale (VAS) scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort.
  This measurement was taken prior to the participant wash-out period
  units on a scale | 69 (20) | 67 (16) | 65 (18) | 67 (18)
Tactile (g) [Mean (Standard Deviation); unit: grams] — The secondary efficacy outcome will be the increase in tactile stimulus force from baseline to 8 weeks. Assessment of Change in tactile sensitivity will be assessed using the Yeaple Electronic Force Sensing Probe.The explorer tip will be applied perpendicular to the tooth surface and a pressure load applied starting at 10 g and increasing to 80g. The load at which the subject says "yes" will be recorded. (Baseline screening will begin at 30g) This measurement was taken prior to washout period.
  grams | 15 (7) | 15 (7) | 16 (7) | 15.3 (7)

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Cold Air Stimulus
Description: The primary efficacy outcome will be the decrease in cold air stimulus sensitivity (VAS score) from baseline to 8 weeks. Assessment of change in cold air sensitivity will be conducted using air delivered from a standard dental unit air syringe at room temperature (~70°F±3°F)(~21°C±2°C) and a pressure of 60psi (± 5psi). Assessment of sensitivity will be carried out using Visual Analog Scale (VAS). Tooth sensitivity was measured using a Cold Air Stimulus. When being assessed, participants rated their perception of the pain/discomfort experienced when cold air was directed at the exposed root of each tooth by marking a single vertical line on a Visual Analogue Scale (VAS) scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort.
Time Frame: Week 0 (baseline), 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Toothpaste 1 | Toothpaste 2 | Toothpaste 3
Number analyzed (Participants) | 62 | 59 | 62
units on a scale
  Week 0 (Baseline) | 71.4 (1.4) | 72.2 (1.47) | 71.9 (1.61)
  Week 4 | 51.1 (1.84) | 51.9 (2.28) | 62 (2)
  Week 8 | 35.6 (1.9) | 37.7 (2.19) | 48.4 (2.21)

2. Secondary Outcome: Measurement of Tactile Stimulus
Description: The secondary efficacy outcome will be the increase in tactile stimulus force from baseline to 8 weeks. Assessment of Change in tactile sensitivity will be assessed using the Yeaple Electronic Force Sensing Probe.The explorer tip will be applied perpendicular to the tooth surface and a pressure load applied starting at 10 g and increasing to 80g. The load at which the subject says "yes" will be recorded. (Baseline screening will begin at 30g).
Time Frame: Week 0 (baseline), 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Toothpaste 1 | Toothpaste 2 | Toothpaste 3
Number analyzed (Participants) | 62 | 59 | 62
Grams
  0 weeks (Baseline) | 13.7 (0.48) | 14.1 (0.57) | 14.8 (0.57)
  4 Weeks | 23.6 (1.15) | 23.2 (1.37) | 17.7 (1.06)
  8 weeks | 31.7 (1.58) | 28.7 (1.77) | 22.9 (1.27)

ADVERSE EVENTS:
Time Frame: Study start to 8 weeks
Description: Adverse events related to study participation were collected.
Arm/Group | Toothpaste 1 | Toothpaste 2 | Toothpaste 3
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/64 | 0/64
Other Adverse Events (participants affected / at risk) | 0/64 | 0/64 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT04590040/Prot_SAP_000.pdf